CLINICAL TRIAL: NCT05971823
Title: Effects of Electronic Cigarette Flavors on Abuse Liability in Smokers (P3-Taste)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20025464; 2U54DA036105 (NIH)
Record Dates: First submitted 2023-07-14; First posted 2023-08-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Electronic Cigarette Use
Keywords: Electronic Cigarette; Nicotine Flux; Tobacco Use
MeSH Terms: conditions — Vaping; Tobacco Use | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Participants will complete 4, within-subject, laboratory sessions that differ by the product used: 1) own brand cigarette, 2) NJOY Ace 2.4% nicotine ECIG (Menthol and Classic Tobacco flavor), 3) NJOY Ace 5.0% nicotine ECIG (Menthol and Classic Tobacco flavor), and 4) NJOY Daily ECIG 6% nicotine (Menthol and Extra Rich Tobacco). The first condition for all participants will be their own brand cigarette. The subsequent three sessions will be assigned using a Latin-square following enrollment, and within each session participants will sample and evaluate two flavors of each session's product (session flavor order is incorporated into the Latin-square condition order assignment).
Who Masked: Participant
Masking Description: Participants will be blinded to device nicotine concentration and flavor used during ECIG sessions. No blinding will occur for the own brand condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Own Brand Cigarette (Active Comparator)
  Interventions: Other: Tobacco product administration and assessment
- NJOY Ace 2.4% nicotine ECIG - Menthol flavor (Experimental)
  Interventions: Other: Tobacco product administration and assessment
- NJOY Ace 2.4% nicotine ECIG - Classic Tobacco flavor (Experimental)
  Interventions: Other: Tobacco product administration and assessment
- NJOY Ace 5.0% nicotine ECIG - Menthol flavor (Experimental)
  Interventions: Other: Tobacco product administration and assessment
- NJOY Ace 5.0% nicotine ECIG - Classic Tobacco flavor (Experimental)
  Interventions: Other: Tobacco product administration and assessment
- NJOY Daily 6.0% nicotine ECIG - Menthol flavor (Experimental)
  Interventions: Other: Tobacco product administration and assessment
- NJOY Daily 6.0% nicotine ECIG - Extra Rich Tobacco flavor (Experimental)
  Interventions: Other: Tobacco product administration and assessment

INTERVENTIONS:
Other: Tobacco product administration and assessment — Subjective measures 1 is followed by product sampling that includes 5 self-directed ECIG/own brand cigarette puffs over 10 minutes. After sampling is complete participants complete subjective measures 2. Ten minutes after their sampling has been completed, they complete subjective measures 3 and the behavioral economic task(s). These activities are preceded and followed by cardiovascular response assessment.

SUMMARY:
The purpose of this study is to determine if abuse liability indices will be impacted by varying flavors and e-cigarette (ECIG) nicotine delivery capability (i.e., nicotine flux) among current combustible cigarette users.

The investigators will compare abuse liability indices between three FDA-authorized ECIG products that vary in nicotine flux (but are all tobacco flavor) and own brand cigarettes. The investigators will also test the influence of ECIG flavor availability (tobacco vs. menthol) within three ECIG product classes.

ELIGIBILITY:
Inclusion Criteria:

* healthy (determined by self-report)
* at least 18 years old
* willing to provide informed consent
* able to attend the lab and use designated products according to study protocol
* smoke cigarettes at least 3 days per week and on those days at least 1 cigarette smoked per day
* positive urine cotinine test

Exclusion Criteria:

* Women if they are breast-feeding or test positive for pregnancy (by urinalysis) at screening.
* Some study details about the eligibility criteria are purposely omitted at this time to preserve scientific integrity. Full details will be posted at the conclusion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Breakpoint of Drug Purchase Task (DPT) | Each DPT will be completed twice per study session, about 55 minutes into the session and again at 120 minutes into the session
  The DPTs will yield measures of willingness to pay and measures of price sensitivity for session-specific tobacco products. Choices made during this task are not reinforced during the session.
Elasticity of Drug Purchase Task (DPT) | Each DPT will be completed twice per study session, about 55 minutes into the session and again at 120 minutes into the session
  The DPTs will yield measures of willingness to pay and measures of price sensitivity for session-specific tobacco products. Choices made during this task are not reinforced during the session.
Omax of Drug Purchase Task (DPT) | A DPT will be Each DPT will be completed twice per study session, about 55 minutes into the session and again at 120 minutes into the session once for each arm.
  The DPTs will yield measures of willingness to pay and measures of price sensitivity for session-specific tobacco products. Choices made during this task are not reinforced during the session.
Pmax of Drug Purchase Task (DPT) | Each DPT will be completed twice per study session, about 55 minutes into the session and again at 120 minutes into the session
  The DPTs will yield measures of willingness to pay and measures of price sensitivity for session-specific tobacco products. Choices made during this task are not reinforced during the session.
Intensity of Drug Purchase Task (DPT) | Each DPT will be completed twice per study session, about 55 minutes into the session and again at 120 minutes into the session
  The DPTs will yield measures of willingness to pay and measures of price sensitivity for session-specific tobacco products. Choices made during this task are not reinforced during the session.
Cross-price elasticity of the Cross Product-DPT | Each CP-DPT will be completed twice per study session, about 55 minutes into the session and again at 120 minutes into the session
  The Cross Product (CP)-DPTs assess cross-product purchasing behaviors between various tobacco products offered at a fixed amount and own brand cigarettes offered at varying prices.

OTHER OUTCOMES:
Subjective measures of nicotine withdrawal | Up to 55 minutes (session 1) and up to 120 minutes (sessions 2-4) into the session
  Nicotine withdrawal will be measured using the Adapted Minnesota Nicotine Withdrawal Scale (MNWS), higher numbers indicate more nicotine dependence.
Subjective measures of nicotine side effects | Up to 55 minutes (session 1) and up to 120 minutes (sessions 2-4) into the session
  Nicotine side effects will be measured using the Direct Effects of Nicotine Scale (DENS), higher scores indicate more intense nicotine side effects.
Subjective measures of product effects | Up to 55 minutes (session 1) and up to 120 minutes (sessions 2-4) into the session
  Product effects will be measured using Direct Effects of Tobacco VAS Scale, higher scores indicate more intense product effects.
General Labeled Magnitude Scale | Up to 55 minutes (session 1) and up to 120 minutes (sessions 2-4) into the session
  Perceptions of electronic cigarette effects will be measured using the General Labeled Magnitude Scale (gLms), higher scores indicate stronger perceptions of nicotine effects.
Labeled Hedonic Scale | Up to 55 minutes (session 1) and up to 120 minutes (sessions 2-4) into the session
  Labeled Hedonic Scale measures nicotine abstinence symptoms, higher scores indicate higher abstinence symptoms
Change in Heart Rate | Recorded throughout each 1 hour and 10 minutes/2 hour and 15 minute study session using automated software every 10 seconds.
  Heart rate (measured in bpm)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline O Cobb, PhD, Principal Investigator — Virginia Commonwealth University; Andrew Barnes, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Center for the Study of Tobacco Products, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT05971823/ICF_000.pdf